CLINICAL TRIAL: NCT03967496
Title: Assessment of Immediate Postoperative Delirium (IPD) in Adult Patients: Incidence, Implication of Type of Anesthesia and Identification of Other Etiological Factors
Brief Title: Assessment of Immediate Postoperative Delirium (IPD) in Adult Patients: Incidence and Etiologic Factors
Acronym: AIPDAP
Status: Completed | Type: Observational
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Sponsor
Other Study IDs: MREC #1829
Record Dates: First submitted 2019-05-19; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Delirium; Anesthesia; Adverse Effect
Keywords: delirium; postoperative complications; anesthesia recovery period
MeSH Terms: conditions — Delirium; Postoperative Complications | interventions — Anesthesia, Conduction; Anesthesia, General; Endoscopy; Laparoscopy; Conversion to Open Surgery; Comorbidity; Hemoglobin, Sickle; Metformin; Lisinopril; Amlodipine; Insulin; Atorvastatin; Hydralazine; Bisoprolol; Leukocyte Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No Delirium: No Delirium: CAM-ICU score of less than 3 throughout Post-Anesthesia Care Unit stay
  Interventions: Procedure: Types of Anesthesia; Procedure: Access of Surgery; Other: Comorbidities; Drug: Preoperative Medication; Diagnostic Test: Routine blood test
- Initial Delirium: Initial Delirium: CAM-ICU score of 3 or more at 15 minutes following end of anesthesia and/or at 30 minutes following end of anesthesia
  Interventions: Procedure: Types of Anesthesia; Procedure: Access of Surgery; Other: Comorbidities; Drug: Preoperative Medication; Diagnostic Test: Routine blood test
- Delirium: Delirium: CAM-ICU score of 3 or more immediately prior to discharge from Post-Anesthesia Care Unit
  Interventions: Procedure: Types of Anesthesia; Procedure: Access of Surgery; Other: Comorbidities; Drug: Preoperative Medication; Diagnostic Test: Routine blood test

INTERVENTIONS:
Procedure: Types of Anesthesia — General Anesthesia includes: Inhalational anesthesia and total intravenous anesthesia.
  Regional blocks includes: Spinal Anesthesia, Epidural Anesthesia, Plexus Block, Peripheral Nerve Block,... etc Monitored Anesthesia Care: No anesthetic administered but care given for hemodynamic and blood sugar control intraoperatively.
  Other Names: Regional Anesthesia; Monitored Anesthesia Care; General Anesthesia
Procedure: Access of Surgery — Type of surgical access
  Other Names: Endoscopy; Laparoscopy; Open surgery
Other: Comorbidities — A patient may have more than one comorbidity
  Other Names: Diabetes; Hypertension; Acute Kidney injury; Chronic Kidney Dysfunction; Ischemic Heart Disease; Bronchial Asthma; Dyslipidemia; Sickle Cell Disease; No Comorbidity
Drug: Preoperative Medication — Preoperative medications
  Other Names: Metformin; Lisinopril; Amlodipine; Insulin; Atorvastatin; Hydralazine; Bisoprolol
Diagnostic Test: Routine blood test — Preoperative and Intraoperative Investigations
  Other Names: Serum hemoglobin; White cell count; Serum sodium; Serum potassium; Serum urea; Serum creatinine; Serum bicarbonate; Serum albumin; Random blood sugar

SUMMARY:
Delirium is considered to be acute failure of central nervous system. It is acute confusional state characterized by decline from baseline mental level, attention deficit and disorganized thinking.

Postoperative delirium is known to prolong length of stay in hospital, cause functional decline and dementia, increase all-cause mortality and increase the medical cost. It is also associated with other outcomes like cardiac arrest, ventricular tachycardia or fibrillation, myocardial infarction, pulmonary edema, pulmonary embolism, bacterial pneumonia, respiratory failure requiring intubation, renal failure requiring dialysis and stroke.

There are well known predisposing and precipitating factors related to its etiology. However, the effect of type of anesthesia is not very clear. There have been no major clinical trials in this part of the world to delineate the incidence of immediate postoperative delirium (IPD). The investigators have undertaken this prospective observational study to determine the incidence of IPD and its etiological factors in adult patients during their stay in the Post-Anesthesia Care Unit (PACU) following surgery under different types of anesthesia (general anesthesia, regional anesthesia and monitored anesthesia care). The study was done over a period of about three months.

Assessment for delirium was done using Confusion Assessment Method-Intensive Care Unit (CAM-ICU score, English/Arabic version). Sedation and Agitation were assessed using Richmond Agitation Sedation Score (RASS). Pain was assessed using Numeric Pain Score (NPS). Assessment was done within 24 hours prior to surgery and was repeated at three different intervals in PACU. Details of perioperative management were recorded and analyzed. The incidence of IPD and its etiologic factors were identified thereby leading to corrective action.

DETAILED DESCRIPTION:
Decision to perform this observational study was made due to the lack of information on the local incidence and risk factors for the development of immediate postoperative delirium (IPD).

A literature review was done to study the already implicated perioperative causative factors as well as other significant perioperative factors.

A consultant neurologist was contacted to confirm the appropriateness of using CAM-ICU, RASS and NPS as assessment tools for the study. Doctors and nurses were trained on the proper use of the assessment tools using educational material at www.icudelirium.org. Permission was obtained from the author who has done validation of arabic version of CAM-ICU score. A proforma was prepared and local Ethical committee approval was obtained.

A pilot study of 24 cases showed the incidence of IPD to be about 25%. The investigators expected to have a total of 600 adult cases undergo anesthesia during the study period of three months. Based on a population size of 600 patients, a level of confidence of 95% and an error of 10% on either side, the optimum sample size was calculated as 395 patients.

The details of the study were explained to each patient with help of information sheet by a dedicated nurse and a doctor well versed in local language. After patient agreement, a written informed consent was obtained. The preoperative scoring of pain, anxiety and agitation and delirium was done by a dedicated nurse under supervision of a doctor who was not involved in providing anesthesia to the patient. Pain was assessed using NPS, sedation/agitation/anxiety using RASS and delirium using CAM-ICU score.

Patient identity was concealed and names were not written in the master chart. The data were entered and identified by the hospital medical registration number (MRN) as well as code number. The patient data were kept locked with password protected file by principal investigators. The premedication choice, anesthetic technique and intraoperative management were carried out in the usual way and recorded on proforma.

Further patient specific data were obtained using the Hospital Information System and Operating Room record. The following data were recorded for each patient:

Demographic Data: Age, gender of the patient

Comorbidity Data: All co-morbidities of patient like diabetes, hypertension, bronchial asthma, ischemic heart disease, jaundice, carcinoma, liver disease, kidney disease, drug addiction, alcoholism, sickle cell disease, medication details and any other co-morbidities.

Laboratory Data: hemoglobin level, creatinine, electrolyte levels, serum albumin, ammonia level and any blood work done preoperative, intraoperative or postoperative in PACU.

Surgical Data: diagnosis, urgency and name of surgery

Peri-operative Anesthetic Data: American Society of Anesthesiologists (ASA) class, premedication, pre-operative medications, hydration status, anesthetic method, analgesics, prophylactic anti-emetic drugs, intraoperative hemodynamic parameters, oxygen saturation, ventilation status, acid-base status, presence of sepsis, fluid and electrolyte imbalance, pain, myocardial infarction, hypo/hyperthermia, alcohol withdrawal and other significant conditions.

Presence of an airway, urinary catheter or a surgical drain at admission to PACU was also recorded.

At the end of anesthesia, all patients were transferred to PACU. The management of the patient was done in the usual manner as prescribed by the involved anesthetist and carried out by allocated PACU nurse. Patients were assessed for pain, agitation, sedation and delirium using NPS, RASS and CAM-ICU score by another trained staff nurse who was not involved in patient management. Scoring was done at fifteen minutes from end of anesthetic, thirty minutes from end of anesthetics and just prior to discharge from PACU (up to 120 minutes from end of anesthetic).

Postoperative course (presence of delirium, requirement of treatment for delirium, length of stay, postoperative complications, admission to high dependency unit or Intensive care unit) was followed via electronic patient record and recorded by concerned anesthetist on the proforma.

The proforma were handed over to the principal investigator and were kept locked. The recorded patient data except the name were entered by one of the assigned co-investigator into the master chart. A copy of master chart without MRN was sent to statistician for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (more than 18 years old) scheduled for Elective and Emergency surgery under anaesthesia.
* Adult patients with ASA- 1 2 or 3 status (American Society of Anaesthesiologists Risk Stratification),
* Patients getting anesthesia: general, regional and monitored anesthesia care.
* Patients undergoing open/laparoscopic/endoscopic surgery.

Exclusion Criteria:

* Refusal to consent
* Patients with ASA- 4 and above risk stratification. Critically ill and unstable patients, shifted from ICU setting and for Emergency surgery.
* Patients with neurological conditions like dementia, psychosis, depression, stroke, head injury and any other pre-existing neurological disease which may interfere with the assessment of delirium.
* Extubation in deep plane of anesthesia where patient is not responsive to verbal commands.
* Deaf and dumb patients
* Inability to comprehend patient language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults undergoing surgery with any type of anesthesia and any type of surgery under ASA grades 1-3, having no prior neurological abnormalities.
Sampling Method: Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Onset of Immediate postoperative delirium (IPD) in adult patients | During PACU stay up to 2 hours.
  Incidence of Immediate postoperative Delirium during Post-Anesthesia-Care-Unit (PACU) stay (at either 15 minutes or 30 minutes after end of anesthesia) as well as at the time of discharge from PACU
Implication of Type of Anesthesia on incidence of Immediate Postoperative Delirium | Intraoperative period
  Includes General Anesthesia (Inhalational as well as Total intravenous anesthesia), Regional Anesthesia and Monitored anesthesia care
Effect of Perioperative risk factors on incidence of Immediate Postoperative Delirium | Perioperative period prior to delirium assessment.
  Perioperative risk factors include: Electrolyte imbalance, anemia, co-morbidities like diabetes, hypertension, ischemic heart disease, chronic kidney diseases etc, preoperative medications like antihypertensives, oral hypoglycemics, insulin, antiplatelets, etc. All details of perioperative management were recorded.

SECONDARY OUTCOMES:
Postoperative Length of stay | Postoperative period up to 8 weeks
  From Day of Surgery till Discharge
Postoperative Complications | Postoperative period up to 8 weeks
  urinary infection, Pneumonia, wound infection, Multi-organ failure or any other complications during that surgical episode.
Mortality rate | Postoperative episode up to 8 weeks
  Mortality due to All causes during the specific postoperative episode up to 8 weeks
Percentage of cases requiring Postoperative Delirium treatment | Postoperative period up to 8 weeks
  Pharmacological as well as Non-pharmacological treatment administered during the postoperative stay in the specific surgical episode up to 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: ALI AL ABADI, MBCHB FRCA, Study Chair — SULTAN QABOOS UNIVERSITY HOSPITAL
Locations (1):
- Sultan Qaboos University Hospital,, Muscat, Oman

IPD SHARING:
Plan to Share IPD: No
As per the Institutional norms we are not supposed to share the data with regards to the study with others.

REFERENCES:
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Neufeld KJ, Leoutsakos JM, Sieber FE, Wanamaker BL, Gibson Chambers JJ, Rao V, Schretlen DJ, Needham DM. Outcomes of early delirium diagnosis after general anesthesia in the elderly. Anesth Analg. 2013 Aug;117(2):471-8. doi: 10.1213/ANE.0b013e3182973650. Epub 2013 Jun 11. PMID 23757476
- [Background] Marcantonio ER, Goldman L, Mangione CM, Ludwig LE, Muraca B, Haslauer CM, Donaldson MC, Whittemore AD, Sugarbaker DJ, Poss R, et al. A clinical prediction rule for delirium after elective noncardiac surgery. JAMA. 1994 Jan 12;271(2):134-9. PMID 8264068
- [Background] Whitlock EL, Vannucci A, Avidan MS. Postoperative delirium. Minerva Anestesiol. 2011 Apr;77(4):448-56. PMID 21483389